CLINICAL TRIAL: NCT07379086
Title: Determinants of Primary Care Health Professionals' Numeracy Skills and Practices and Association With Patient Health Literacy and Quality of Care
Acronym: Num-Pro-Qual
Status: Not yet recruiting | Type: Observational
Sponsor: MSPU de Pins-Justaret (Other)
Responsible Party: Sponsor
Other Study IDs: Num-Pro-Qual
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Health Literacy; Numeracy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To enable appropriate risk representation for patients, health care professionals (HCPs) must have a personal understanding of quantitative data. To date, a limited number of studies on physicians' numeracy skills and practices show that, although physicians perform better than the general population, not all physicians have mastered basic numeracy skills. Low numeracy among physicians was associated with lower quality adherence to good practice recommendations, inaccurate inferences about test results and side effect risks, and reluctance to share numerical information with patients. The primary objective will be to explore the determinants of the objective numeracy level of primary care professionals. A cross-sectional survey will be conducted on a sample of primary care professionals practicing in the west of Occitanie (former Midi-Pyrenées region). Objective numeracy will be measured using the Adaptive Berlin Numeracy Test (ABNT) and the Abbreviated Numeracy Scale, whereas subjective numeracy will be assessed using the Subjective Numeracy Scale (SNS-3). The Health Literacy Questionnaire (HLQ) will be used for patients.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years of age
* having declared one of the participating general practitioners as their treating physician
* declaring to be regularly followed by one of the participating physicians (at least 2 consultations in the last 12 months) for whom a non-opposition collection was carried out

Exclusion criteria:

* diagnosis of major cognitive impairment
* lack of mastery of the French language or lack of ability to understand oral or written instructions
* patient under legal protection regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Objective numeracy | Baseline
  Objective numeracy, as measured by the Adaptive Berlin Numeracy Test (ABNT)